CLINICAL TRIAL: NCT01271101
Title: The Efficacy and Safety of Anticoagulation in Chinese Patients With Non-ST Segment Elevation Acute Coronary Syndrome
Acronym: EASY-CHINA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Jinming Yu, School of Public Health, Fudan University
Other Study IDs: EASY-CHINA
Record Dates: First submitted 2011-01-05; First posted 2011-01-06 (Estimated); Last update posted 2011-01-06 (Estimated); Status verified 2010-07

CONDITIONS: Acute Coronary Syndrome
Keywords: Non-ST-elevated acute coronary syndromes (NSTE-ACS); anticoagulation
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- anticoagulant

SUMMARY:
The primary objective of the EASY-CHINA Registry is to describe the clinical epidemiology of Chinese patients with NSTE-ACS, to evaluate their current anticoagulation management in China, and the resources used for it.

DETAILED DESCRIPTION:
Non-ST-elevated acute coronary syndromes (NSTE-ACS)are the leading cause of emergency medical care in the USA. In China, these syndromes have also become the major causes of morbidity and mortality and account for several thousands of death and hospitalizations annually. Anti-platelet drugs, anticoagulants and intervention therapy for high-risk NSTE-ACS patients may increase bleeding events while reducing ischemic coronary events. There are some evidences supporting the association between hemorrhagic complications and short- and long-term mortality. Therefore, future advances in antithrombotic therapy for NSTE-ACS need to focus on reducing ischemic event rates without increasing hemorrhagic complication rates. In this general framework, there is the need for an appropriate adoption of the available evidences concerning therapeutic strategies, specifically the use of the different antithrombotic strategies, in real world patients in order to further improve their outcomes.The primary objective of this study is to describe the clinical epidemiology of Chinese patients with NSTE-ACS, and to evaluate their current management in China. This study will be an observational survey, thus zero interference is emphasized throughout it. No randomization, blinding or special treatment will be assigned for the subjects. Issues concerning the care of subjects are completely left to the discretion of investigators in order to collect the real-world information about the pharmacological treatments for NSTE-ACS patients in china.

ELIGIBILITY:
Inclusion Criteria:

* with symptoms of UA or MI without persistent ST elevation and at least 1 of the following additional criterias: 1)troponin T or I or CK-MB above the upper limit of normal,2)electrocardiogram (ECG) changes compatible with ischemia (ie, ST depression at least 1mm in 2 contiguous leads or T-wave inversion >3 mm),3)any dynamic ST shift or transient ST elevation
* Must be willing to signed informed consent
* age from 21-80 years
* without pregnancy or under contraception

Exclusion Criteria:

* age<20 or >80 years
* any contraindication to anticoagulant
* hemorrhagic stroke within 12 months
* indication for anticoagulation other than ACS
* prior enrollment in anticoagulants trials in ACS
* revascularization procedure performed for the qualifying event in one month
* severe renal insufficiency (ie,serum creatinine>=3 mg/dL or 265umol/L)
* pregnancy or breast-feeding women
* life expectancy<6 months
* enrollment in other medicine trials in 3 months
* with mental illness or uncooperative

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chinese patients with non-ST-elevated acute coronary syndrome
Sampling Method: Non-Probability Sample
Enrollment: 1800 (Estimated)
Dates: Start 2010-07; Primary Completion 2011-03 (Estimated); Study Completion 2011-08 (Estimated)

PRIMARY OUTCOMES:
the composite of death, MI, refractory ischemia, or stroke and the major bleeding | 9 days

SECONDARY OUTCOMES:
the composite of death, MI, refractory ischemia, or stroke | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Jinming Yu, Doctor, Principal Investigator — School of Public Health，Fudan University
Locations (1):
- School of Public Health, Fudan University, Shanghai, Shanghai Municipality, China